CLINICAL TRIAL: NCT04728477
Title: Accuracy, Precision and Trending Abilities of Novel Optical Smartphone Application for Blood Pressure Measurements in Critically Ill Patients: A Method Comparison Study Against the Arterial Line as the Reference Method
Brief Title: Evaluation of Novel Optical Smartphone Application for Blood Pressure Measurements in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Study Director, Erasme University Hospital
Other Study IDs: P2020/665
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OPti BP measurements — measurement of blood pressure with the new smartphone App ( OPTIBP)

SUMMARY:
Evaluation of a novel mobile application designed to estimate blood pressure (systolic-diastolic and mean arterial pressure) based on collected optical signals on patient's finger treated in intensive care unit patients

DETAILED DESCRIPTION:
The purpose of the study is to compare the blood pressure values measured by a novel mobile phone application ( camera of the smartphone will be obstructed by the patient's right index) and the values measured by reference method used (the radial arterial line)

All patients admitted in the intensive care unit at Erasme Hospital Brussels, Belgium will be recruited and if they have an arterial line for at least two days

The OptiBP Application is a mobile application installed on a mobile phone which is a non-invasive data-logger intended to acquire physiological data from patients. By applying the patient's finger on a smartphone's camera, a movie is generated and transformed into values of diastolic, mean and systolic blood pressure.

Three measures will be taken (spaced by one minute) with both methods each hour for 5 hours and this will be done for 2 days.

The patient's blood pressure will be measured in parallel with the mobile application and with the reference equipment (arterial line).

Then, the values obtained by the two methods will be compared to confirm the reliability of the data obtained with the novel mobile application.

The goal is therefore to compare blood pressure values as obtained by the analysis of the data recorded by the OptiBP Mobile Application, against simultaneous measurements provided by the arterial line (gold standard)

ELIGIBILITY:
Inclusion Criteria:

* All Intensive care unit patients with an arterial catheter for at least 48 hours
* Informed Consent as documented by signature

Exclusion Criteria:

* Patients or families that cannot sign informed consent
* Patients in emergency situation, and unstable
* Dyshythmia like bigeminy, trigeminy, isolated Ventricular Premature Beats (VPB), atrial fibrillation
* Lesion or deficiency on hand, preventing index obstruction of smartphone's camera
* Known contact dermatitis to nickel/chromium

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All intensive care unit patients with an arterial catheter for at least 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of blood pressure between the new smartphone App and the radial arterial line | 48 hours
  Comparative blood pressure measurement with the investigational device and the invasive reference method (arterial line).

SECONDARY OUTCOMES:
Usability assessment | at 48 hour
  Identification of possible use error in the manipulation of the device and in the performance of the measure

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre JOOSTEN, MD PhD, Principal Investigator — ERASME
Locations (1):
- ERASME, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desebbe O, Anas C, Alexander B, Kouz K, Knebel JF, Schoettker P, Creteur J, Vincent JL, Joosten A. Evaluation of a novel optical smartphone blood pressure application: a method comparison study against invasive arterial blood pressure monitoring in intensive care unit patients. BMC Anesthesiol. 2022 Aug 15;22(1):259. doi: 10.1186/s12871-022-01797-0. PMID 35971072